CLINICAL TRIAL: NCT01269489
Title: Health-related Quality of Life in General Slovenian Poplation Assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Core Quality-of-Life Questionnaire QLQ-C30
Brief Title: Health-related Quality of Life in General Slovenian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Vaneja Velenik, PhD, MD, Institute of Oncology
Other Study IDs: 134/09/09
Record Dates: First submitted 2011-01-01; First posted 2011-01-04 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Health-related Quality of Life
Keywords: quality of life; general Slovenian population; EORTC QLQ C30

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- general population: a representative sample from general Slovenian population

SUMMARY:
The purpose of the study is to obtain reference data on health-related quality of life for the functional and symptom scales and single items of the European Organisation for Research and Treatment of Cancer Core Quality-of-Life Questionnaire (EORTC QLQ C30) in a representative sample of Slovenian general population.

DETAILED DESCRIPTION:
A sample of at least 600 people from the Slovenian population, randomly selected, age 18 years and more, representing geografic diversity, will take part in this postal survey. The EORTC QLQ C30 and a questionnaire about demografic data will be send by mail. This is the first study to obtain reference data from the EORTC QLQ C30 in a sample from the general Slovenian population. The results will serve as guidelines for interpreting health-related quality-of-life of different groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 y and more

Exclusion Criteria:

* serious comorbidity
* previously treated for cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: sample from general Slovenian population
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vaneja Velenik, PhD, MD, Principal Investigator — Institute of Oncology Ljubljana Slovenia
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia

REFERENCES:
- [Background] Cocks K, King MT, Velikova G, Fayers PM, Brown JM. Quality, interpretation and presentation of European Organisation for Research and Treatment of Cancer quality of life questionnaire core 30 data in randomised controlled trials. Eur J Cancer. 2008 Sep;44(13):1793-8. doi: 10.1016/j.ejca.2008.05.008. Epub 2008 Jul 1. PMID 18599286
- [Background] Fayers P, Bottomley A; EORTC Quality of Life Group; Quality of Life Unit. Quality of life research within the EORTC-the EORTC QLQ-C30. European Organisation for Research and Treatment of Cancer. Eur J Cancer. 2002 Mar;38 Suppl 4:S125-33. doi: 10.1016/s0959-8049(01)00448-8. PMID 11858978